CLINICAL TRIAL: NCT03389256
Title: A Randomized, Controlled Phase II Clinical Trial of Apatinib in Combination With EGFR-TKI Versus EGFR-TKI for Non-squamous, Non-small Cell Lung Cancer(NSCLC) With T790M-negative After the Failure of EGFR-TKI Therapy
Brief Title: Apatinib in the Treatment of Patients With EGFR T790M-Negative NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Juan LI, MD, MD, Sichuan Cancer Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APTN-NSCLC-201712
Record Dates: First submitted 2017-12-26; First posted 2018-01-03 (Actual); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms; Non-Small-Cell Lung
Keywords: apatinib; T790 negative; NSCLC
MeSH Terms: conditions — Lung Diseases; Neoplasms; Respiratory Tract Diseases; Thoracic Neoplasms | interventions — apatinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib combine with EGFR-TKI (Experimental): Every 4 weeks 1 cycle, evaluated the efficacy and safety once every 2 cycles, treat until disease progression or intolerable toxicity
  Interventions: Drug: Apatinib; Drug: EGFR-TKI
- EGFR-TKI (Active Comparator): Every 4 weeks 1 cycle, evaluated the efficacy and safety once every 2 cycles, treat until disease progression or intolerable toxicity
  Interventions: Drug: EGFR-TKI

INTERVENTIONS:
Drug: Apatinib — Apatinib mesylate tablets 250 mg qd po, if the patient can tolerate the toxic side effects, adjust the dose to 500mg qd po after 1 week.
  Other Names: apatinib tablets
  Arms: apatinib combine with EGFR-TKI
Drug: EGFR-TKI — Imatinib tablets, 125 mg tid po; gefitinib tablets, 250 mg qd po; erlotinib tablets, 150 mg qd po
  Other Names: Imatinib、Gefitinib or Erlotinib

SUMMARY:
This phase 2 study is designed to evaluate the safety and activity of apatinib,a tyrosine kinase inhibitor that selectively inhibits the vascular endothelial growth factor receptor-2, in combination with EGFR-TKI in NSCLC with T790M-negative after the failure of EGFR-TKI therapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed stage IIIB, IV non-squamous non-small cell lung cancer, with measurable lesions (the long axis of tumor lesions ≥ 10mm with CT, the short axis of lymph node lesions ≥ 15mm with CT, the lesions not receive radiotherapy, frozen or other local treatment);
* Patients with slow progression on first-line EGFR TKI(erlotinib / icotinib / gefitinib) treatment;
* No T790M mutation including an assessment from tumor biopsy obtained while on or subsequent to the most recent EGFR TKI therapy;
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2;
* Life expectancy of more than 3 months;
* Adequate bone marrow function: WBC ≥ 3.0 ×10 E+9/L, neutrophil ≥ 1.5 × 10 E+9/L, platelets ≥ 80 × 10E+9/L,Hb ≥ 10.0g/dL;a total bilirubin (TBil) of ≤1.5 upper normal limitation (UNL), a alanine aminotransferase (ALAT) and aspartate aminotransferase (ASAT) of ≤3UNL or ≤5UNL in case of liver metastasis, a creatinine (Cr) of ≤ 1.5 UNL; a creatinine clearance rate ≥ 50ml/min (Cockcroft-Gault);
* Female subjects of child-bearing potential must agree to use contraceptive measures starting 1 week before the administration of the first dose of apatinib until 8 weeks after discontinuing study drug. Male subjects must agree to use contraceptive measures during the study and 8 weeks after last dose of study drug;
* the participants volunteered to join this study should sign the informed consent forms, have better compliance in the follow-up;

Exclusion Criteria:

* Squamous cell carcinoma (including adenosquamous carcinoma); Small cell lung carcinoma (including small cell carcinoma and non-small cell mixed lung carcinoma);
* Active brain metastases, cancerous meningitis, patients with spinal cord compression;
* Rapid progression of the disease or cancer invades vital organs;
* The distance between the tumor lesion and the large blood vessel is less than 5 mm, or there is a central tumor invading local macrovascular;
* obvious pulmonary cavity or tumor necrosis;
* Uncontrollable high blood pressure;
* Grade Ⅱ or above myocardial ischemia or myocardial infarction or arrhythmia control is not good,Ⅲ ~ Ⅳ grade cardiac insufficiency, or cardiac ultrasonography showed left ventricular ejection fraction (LVEF) <50% according to the NYHA standard;
* Have a history of interstitial lung disease or patients with interstitial lung disease;
* Coagulation abnormalities (INR> 1.5 or PT> ULN + 4s or APTT> 1.5 ULN) with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
* There was significant hemoptysis within 2 months prior to enrollment, or a daily hemoptysis volume is 2.5 ml or above;
* A clinically significant bleeding symptom or bleeding tendencies such as gastrointestinal bleeding, hemorrhagic gastric ulcer, fecal occult blood ++ and above, or vasculitis that occurred within 3 months prior to enrollment;
* Aneurysm / venous thrombotic events such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism;
* Arterial / venous thrombotic events such as cerebrovascular accidents (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism within 12 months prior to enrollment;
* Hereditary or acquired bleeding and thrombophilia, such as hemophilia, coagulopathy, thrombocytopenia, hypersplenism；
* Long-term unhealed wounds or fractures;
* Major surgery or severe traumatic injury, fracture or ulcer within 4 weeks prior to enrollment;
* Unable to swallow, chronic diarrhea or intestinal obstruction;
* Abdominal fistula, gastrointestinal perforation or abdominal abscess within 6 months prior to enrollment;
* Urinary protein ≥ ++, 24-hour urinary protein ≥ 1.0 g;
* Active infections require antimicrobial treatment;
* ALK gene abnormalities (gene fusion or mutation occurred);
* Pregnant or lactating women, or women unwilling or unable to take effective contraception;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-12-30 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | up to 24 months
  the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  The length of time from either the date of diagnosis or the start of treatment that half of the patients in a group of patients diagnosed with the disease are still alive.
Duration of response (DOR) | up to 24 months
  From first response to the date of first documented disease progression
Disease Control Rate (DCR) | 24 weeks
  the proportion of patients with a best overall response of CR, PR or SD in the whole body, as assessed per RECIST 1.1 by the investigator.
Overall response rate (ORR) | 24 weeks
  the proportion of patients with a best overall confirmed response of CR or PR in the whole body as assessed per RECIST 1.1 by the investigator
the quality of life (QoL) | up to 36 months
  Analysis of changes from baseline using the quality of life (QoL) instrument

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided